CLINICAL TRIAL: NCT03964649
Title: Comparative Analysis of Outcomes Among Rheumatoid Arthritis Patients Treated With Xeljanz Versus Biologic DMARDs Using a United States Healthcare Claims Database
Brief Title: Comparative Analysis of Outcomes Among Patients Treated With Xeljanz vs Biologics
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921305
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Truven Health MarketScan Research Database: To compare RA-related costs among patients treated with tofacitinib (IR, XR and combined groups) to patients treated with each of the bDMARDs (individually, as well as to TNFi and to non-TNFi each combined as groups).

SUMMARY:
To compare rheumatoid arthritis (RA) patient characteristics, adherence, and costs between patients treated with tofacitinib (IR, XR and combined groups) to patients treated with each of the bDMARDs.

ELIGIBILITY:
Inclusion Criteria:

* At least one claim for methotrexate during the variable-length pre-index period.
* At least one claim for tofacitinib or bDMARDs between 01 February 2016 and 31 July 2019 (the identification period).

Exclusion Criteria:

* Patients with claims for other conditions for which bDMARDs are used during the one-year pre-index period or on the index date: ankylosing spondylitis, Crohn's disease, psoriasis, psoriatic arthritis, or ulcerative colitis will be excluded from the study.
* Patients with evidence of the index medication during the one-year pre-index period will be removed from the analysis. Patients will be allowed to have been treated with (other) bDMARDs during the one-year pre-index period.
* Patients with more than 1 bDMARD or bDMARD with tofacitinib filled on the index date will be removed from the study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will utilize the de-identified claims data in the Truven Health MarketScan Research Database.
Sampling Method: Non-Probability Sample
Enrollment: 7308 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with rheumatoid arthritis (RA), who newly initiated tofacitinib or biologic disease-modifying antirheumatic drug (bDMARDs), between 01 February 2016 and 31 July 2019 (identification period), were identified using Truven Health MarketScan Research database. Data for eligible participants from database were evaluated in this retrospective observational study. Index date = date of first claim for index medication (bDMARDs or tofacitinib) during identification period of 3.5 years.
Pre-assignment Details: Baseline characteristics- age, sex, region of enrollment were evaluated at index date. Other study specific characteristics were observed over 12 months before index date (12 months pre-index baseline period) and/or over variable-length pre-index baseline period. Variable-length pre-index baseline period was minimum of 1 year and could have been maximum up to 5.68 years before index date.
Groups:
- Tofacitinib XR: Participants who started treatment with modified-release (XR) tofacitinib during identification period were included in this arm.
- Tofacitinib IR: Participants who started treatment with immediate-release (IR) tofacitinib during identification period were included in this arm.
- Adalimumab: Participants who started treatment with adalimumab (tumor-necrosis factor-alpha inhibitor [TNFI]) during identification period were included in this arm.
- Certolizumab Pegol: Participants who started treatment with certolizumab pegol (TNFI) during identification period were included in this arm.
- Etanercept: Participants who started treatment with etanercept (TNFI) during identification period were included in this arm.
- Infliximab: Participants who started treatment with infliximab (TNFI) during identification period were included in this arm.
- Golimumab: Participants who started treatment with golimumab (TNFI) during identification period were included in this arm.
- Rituximab: Participants who started treatment with rituximab (non-TNFI) during identification period were included in this arm.
- Tocilizumab: Participants who started treatment with tocilizumab (non-TNFI) during identification period were included in this arm.
- Abatacept: Participants who started treatment with abatacept (non-TNFI) during identification period were included in this arm.
Period: Overall Study
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Started | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Completed | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept | Total
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533 | 7308
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.48 (11.04) | 55.93 (11.26) | 51.42 (10.35) | 56.70 (14.90) | 51.85 (10.89) | 55.85 (12.33) | 55.63 (12.55) | 56.13 (11.90) | 55.99 (11.65) | 55.88 (11.45) | 53.14 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 250 | 2124 | 156 | 1523 | 279 | 302 | 257 | 158 | 448 | 5779
  Male | 67 | 54 | 604 | 36 | 425 | 70 | 74 | 68 | 46 | 85 | 1529
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast Region | 96 | 69 | 422 | 45 | 331 | 51 | 55 | 57 | 41 | 114 | 1281
  United States: North Central Region | 62 | 58 | 605 | 21 | 390 | 74 | 46 | 77 | 37 | 93 | 1463
  United States: South Region | 143 | 137 | 1349 | 104 | 952 | 178 | 235 | 120 | 97 | 256 | 3571
  United States: West Region | 45 | 40 | 348 | 22 | 274 | 46 | 37 | 71 | 29 | 70 | 982
  United States: Unknown Region | 3 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 11
Mean Number of bDMARDs Received During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: number of bDMARDs] — bDMARDs included: Tumor-necrosis factor-alpha inhibitors (TNFi) [adalimumab, etanercept, certolizumab pegol, golimumab, infliximab] and non-TNFi's [abatacept, rituximab and tocilizumab].
  number of bDMARDs | 1.11 (0.32) | 1.40 (0.59) | 1.11 (0.31) | 1.31 (0.80) | 1.06 (0.24) | 1.41 (0.56) | 1.19 (0.45) | 1.31 (0.62) | 1.20 (0.45) | 1.22 (0.42) | 1.23 (0.49)
Mean Number of bDMARDs Received During Variable Length Pre-Index Baseline Period [Mean (Standard Deviation); unit: number of bDMARDs] — Biologic DMARDs included: Tumor-necrosis factor-alpha inhibitors (TNFi) [adalimumab, etanercept, certolizumab pegol, golimumab, infliximab] and non-TNFi's [abatacept, rituximab and tocilizumab].
  number of bDMARDs | 1.46 (0.73) | 1.61 (0.81) | 1.24 (0.55) | 1.88 (1.12) | 1.23 (0.65) | 1.83 (1.09) | 1.58 (0.91) | 1.78 (1.14) | 1.79 (0.95) | 1.58 (0.78) | 1.55 (0.87)
Mean Number of csDMARDs Received During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: csDMARDs] — In this baseline measure mean of number of conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) used during 12 months pre-index period is reported.
  csDMARDs | 1.58 (0.66) | 1.48 (0.66) | 1.56 (0.69) | 1.39 (0.59) | 1.61 (0.72) | 1.56 (0.72) | 1.50 (0.67) | 1.56 (0.68) | 1.49 (0.69) | 1.63 (0.73) | 1.57 (0.70)
Mean Number of csDMARDs Received During Variable Length Pre-Index Baseline Period [Mean (Standard Deviation); unit: csDMARDs] — In this baseline measure mean of number of conventional synthetic disease-modifying antirheumatic drugs (csDMARDs) used during the variable length pre-index period is reported.
  csDMARDs | 1.91 (0.89) | 1.88 (0.87) | 1.76 (0.82) | 1.66 (0.80) | 1.82 (0.85) | 1.76 (0.86) | 1.73 (0.82) | 1.93 (0.91) | 1.71 (0.88) | 2.02 (0.92) | 1.81 (7,308)
Quan-Charlson Comorbidity Score During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: units on a scale] — The mean Quan-Charlson Comorbidity score during pre-index baseline period is reported. Quan-Charlson Comorbidity score predicts probability of death within one year in participants and was based on presence of any diagnosis codes on medical claims at any time during the 12-months pre-index baseline period, based on the international classification of diseases (ICD) diagnosis codes. Total score ranges from 0 to 9.0. A score of 0 indicated that no comorbidities were found. The higher the score, the more likely predicted outcome could result in mortality or higher healthcare resource utilization.
  units on a scale | 1.77 (1.14) | 1.89 (1.32) | 1.63 (1.04) | 1.95 (1.46) | 1.70 (1.13) | 1.94 (1.43) | 1.72 (1.22) | 2.54 (1.81) | 2.01 (1.52) | 2.10 (1.46) | 1.78 (1.23)
Number of Participants With Most Commonly Used Medications During 12 Month Pre-index Baseline Period [Count of Participants; unit: Participants] — Number of participants for each of the most commonly used medications during the 12 months pre-index baseline period are reported.
  Participants
    Methotrexate Sodium | 279 | 220 | 2440 | 155 | 1,732 | 306 | 313 | 253 | 152 | 396 | 6246
    Folic Acid | 226 | 177 | 2,024 | 126 | 1,435 | 230 | 272 | 197 | 122 | 329 | 5138
    Prednisone | 219 | 203 | 1,930 | 123 | 1,379 | 250 | 251 | 232 | 157 | 368 | 5112
    Hydroxychloroquine Sulfate | 106 | 98 | 919 | 43 | 711 | 102 | 109 | 112 | 59 | 211 | 2470
    Acetaminophen/Hydrocodone Bitartrate | 82 | 89 | 768 | 60 | 518 | 122 | 114 | 107 | 75 | 157 | 2092
    Methylprednisolone | 79 | 61 | 684 | 38 | 503 | 81 | 89 | 52 | 39 | 112 | 1738
    Tramadol Hydrochloride | 58 | 64 | 604 | 37 | 462 | 79 | 89 | 84 | 44 | 124 | 1645
    Azithromycin | 89 | 64 | 592 | 50 | 430 | 74 | 94 | 67 | 38 | 126 | 1624
    Meloxicam | 59 | 47 | 647 | 29 | 448 | 73 | 81 | 41 | 36 | 89 | 1550
    Levothyroxine Sodium | 67 | 55 | 498 | 35 | 363 | 65 | 73 | 62 | 43 | 119 | 1380
    Gabapentin | 52 | 34 | 373 | 31 | 315 | 64 | 64 | 53 | 37 | 114 | 1137
    Omeprazole | 42 | 50 | 367 | 22 | 320 | 62 | 62 | 67 | 40 | 92 | 1124
    Albuterol Sulfate | 52 | 48 | 411 | 25 | 282 | 54 | 42 | 47 | 36 | 92 | 1089
    Diclofenac Sodium | 47 | 42 | 410 | 27 | 294 | 62 | 64 | 34 | 28 | 77 | 1085
    Leflunomide | 56 | 50 | 356 | 27 | 283 | 60 | 62 | 44 | 27 | 94 | 1059
    Amoxicillin | 52 | 41 | 365 | 25 | 286 | 47 | 62 | 47 | 29 | 94 | 1048
    Cyclobenzaprine Hydrochloride | 46 | 43 | 367 | 25 | 286 | 45 | 55 | 40 | 35 | 73 | 1015
    Fluticasone Propionate | 55 | 51 | 329 | 29 | 259 | 51 | 46 | 47 | 25 | 70 | 962
    Amoxicillin/Clavulanate Potassium | 60 | 34 | 380 | 19 | 228 | 52 | 36 | 40 | 28 | 80 | 957
    Acetaminophen/Oxycodone Hydrochloride | 40 | 39 | 294 | 23 | 229 | 56 | 41 | 49 | 32 | 82 | 885
    Ibuprofen | 36 | 40 | 318 | 20 | 233 | 59 | 50 | 29 | 27 | 62 | 874
    Ergocalciferol | 48 | 32 | 322 | 25 | 206 | 40 | 56 | 36 | 28 | 60 | 853
    Duloxetine Hydrochloride | 36 | 34 | 289 | 22 | 222 | 47 | 51 | 30 | 28 | 75 | 834
    Ciprofloxacin Hydrochloride | 40 | 38 | 249 | 16 | 219 | 41 | 42 | 52 | 23 | 80 | 800
    Atorvastatin Calcium | 54 | 26 | 285 | 20 | 190 | 51 | 41 | 33 | 29 | 64 | 793
Number of Participants Who Used Opioids or NSAIDs During 12 Months Pre-Index Baseline Period [Count of Participants; unit: Participants] — Number of participants who used at least one opioid or NSAID during pre-index period are reported.
  Participants | 214 | 236 | 1,867 | 134 | 1,360 | 265 | 277 | 229 | 157 | 380 | 5119
Mean Number of Pharmacy Claims for Opioids and NSAIDS During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: pharmacy claims] — The mean number of pharmacy claims for opioids and NSAIDs during the pre-index period are reported. A pharmacy claim was defined as a claim made by participants to their insurance provider in purchasing opioids and NSAIDs from the pharmacy. Population: Here, "overall number of participants analyzed" signifies participants evaluable for this baseline measure.
  pharmacy claims
    number analyzed (Participants) | 214 | 236 | 1867 | 134 | 1360 | 265 | 277 | 229 | 157 | 380 | 5119
    (all) | 4.04 (6.39) | 5.31 (6.85) | 4.08 (5.84) | 4.15 (6.09) | 4.45 (5.80) | 4.84 (5.92) | 4.46 (5.38) | 4.14 (5.23) | 5.05 (6.21) | 4.58 (5.94) | 4.35 (5.89)
Number of Participants Who Used Oral Corticosteroids During 12 Months Pre-Index Baseline Period [Count of Participants; unit: Participants] | 254 | 222 | 2,138 | 134 | 1,515 | 276 | 280 | 249 | 167 | 400 | 5635
Mean Number of Visits to Rheumatologist During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: visits] — In this baseline measure mean of number of visits made by participants to rheumatologist during 12 months pre-index period is reported.
  visits | 4.53 (2.38) | 4.92 (2.90) | 4.65 (2.47) | 5.26 (2.88) | 4.76 (2.62) | 5.60 (2.88) | 5.89 (3.59) | 5.41 (3.06) | 5.79 (3.94) | 5.92 (4.19) | 4.97 (2.89)
Mean Number of Visits to Rheumatologist During Variable-Length Pre-Index Baseline Period [Mean (Standard Deviation); unit: visits] — In this baseline measure mean of number of visits made by participants to rheumatologist during variable length pre-index period is reported.
  visits | 11.28 (8.45) | 12.12 (8.56) | 8.21 (5.98) | 11.43 (9.51) | 8.39 (6.03) | 10.79 (7.79) | 11.25 (8.36) | 13.01 (9.69) | 13.75 (11.80) | 12.43 (8.90) | 9.61 (7.45)
Disease Duration During Variable-Length Pre-Index Baseline Period [Mean (Standard Deviation); unit: days] — Disease duration was defined as the number of days from the first recorded date of diagnosis of rheumatoid arthritis to the date of the index day.
  days | 882.61 (558.81) | 919.71 (437.63) | 570.38 (481.35) | 730.28 (536.06) | 568.98 (474.54) | 661.66 (513.64) | 651.11 (482.93) | 888.34 (541.51) | 806.50 (527.20) | 789.95 (498.75) | 648.91 (504.69)
Out of Pocket Health Care Costs for Healthcare Services During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: dollars] — In this baseline measure out of pocket medical care expenses not reimbursed by insurance during 12 months pre-index period is reported.
  dollars | 1803.44 (1789.99) | 2154.86 (1828.01) | 2152.95 (1741.99) | 2013.10 (1714.01) | 2251.93 (1800.59) | 2287.63 (2494.77) | 2174.31 (1782.74) | 2797.43 (2975.36) | 2174.18 (1553.37) | 2453.28 (2389.53) | 2217.74 (1931.29)
Out of Pocket Health Care Costs for Healthcare Services During Variable Length Pre-Index Period [Mean (Standard Deviation); unit: dollars] — In this baseline measure out of pocket medical care expenses not reimbursed by insurance during variable length pre-index period is reported.
  dollars | 6626.03 (5819.96) | 6549.23 (4717.18) | 6270.02 (5087.71) | 6453.01 (5204.02) | 6510.77 (5550.34) | 6856.14 (6946.33) | 6841.01 (6423.20) | 8934.99 (12740.35) | 7331.39 (5037.30) | 7636.47 (6096.75) | 6672.79 (6042.90)
Number of Participants With Comorbidities of Interest During 12 Months Pre-Index Baseline Period [Count of Participants; unit: Participants] — The comorbidities of interest included cardiovascular diseases, chronic obstructive pulmonary disorder (COPD), asthma, kidney disease, diabetes, depression, anxiety, liver disease, sleep disorders, hypertension, hyperlipidemia. A participant could have greater than (>) 1 comorbidity of interest. Pre-index baseline period was the 12 month duration before the index date. The index date was the date of the first claim for bDMARDs or tofacitinib during the identification period.
  Participants
    Cardiovascular disease | 198 | 189 | 1315 | 110 | 992 | 205 | 208 | 210 | 133 | 328 | 3888
    COPD | 33 | 33 | 248 | 23 | 188 | 46 | 38 | 47 | 34 | 74 | 764
    Asthma | 35 | 38 | 272 | 16 | 210 | 45 | 30 | 35 | 26 | 71 | 778
    Kidney disease | 37 | 30 | 257 | 27 | 192 | 38 | 43 | 55 | 30 | 81 | 790
    Diabetes | 54 | 54 | 424 | 33 | 283 | 65 | 56 | 62 | 33 | 114 | 1178
    Depression | 54 | 58 | 450 | 30 | 376 | 60 | 67 | 58 | 35 | 117 | 1305
    Anxiety | 59 | 57 | 412 | 32 | 343 | 60 | 58 | 50 | 18 | 98 | 1187
    Liver disease | 18 | 17 | 143 | 17 | 111 | 24 | 19 | 31 | 19 | 41 | 440
    Sleep disorders | 44 | 31 | 307 | 18 | 209 | 45 | 49 | 34 | 26 | 79 | 842
    Hypertension | 157 | 153 | 1053 | 96 | 790 | 169 | 172 | 158 | 104 | 268 | 3120
    Hyperlipidemia | 150 | 120 | 931 | 73 | 682 | 155 | 147 | 115 | 88 | 223 | 2684
All cause Inpatient, Outpatient and Emergency Room Visits Costs During 12 Months Pre-Index Period [Mean (Standard Deviation); unit: dollars] — All cause inpatient visit costs consisted of expenses during hospital visit for formal admission. Outpatient visit costs consisted of expenses when participants visited hospital but not for formal admission. Emergency room (ER) visit costs consisted of expenses during visit to hospital emergency room.
  dollars
    Inpatient visits costs | 6,439.48 (24,897.59) | 5,918.18 (31,820.77) | 2796.16 (13970.41) | 5745.63 (21990.52) | 2908.83 (13624.11) | 2802.86 (9813.21) | 5593.85 (28885.69) | 10287.84 (32246.91) | 9475.99 (32796.53) | 4661.57 (16089.35) | 4007.49 (18785.55)
    Outpatient visits costs | 11,764.03 (27,775.60) | 12,056.68 (19,456.56) | 8235.49 (14916.40) | 10585.64 (13522.28) | 8989.76 (18037.61) | 13625.70 (23,398.43) | 11200.01 (20002.68) | 25746.57 (46437.00) | 15879.61 (26952.93) | 14260.86 (19512.63) | 10667.28 (20794.73)
    Emergency Room visits costs | 1,308.81 (3,867.67) | 1,404.59 (5,254.09) | 968.34 (3245.47) | 1035.11 (3080.83) | 1094.48 (3219.72) | 1528.22 (3716.98) | 1014.59 (2993.84) | 1,519.68 (3770.18) | 1721.96 (5667.52) | 1413.05 (4290.22) | 1145.23 (3581.14)
RA Related Inpatient, Outpatient and ER Visits Costs During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: dollars] — RA related inpatient visit costs consisted of expenses during hospital visits for formal admission for RA. Outpatient visit costs consisted of expenses when participants visited hospital but not for formal admission for RA. ER visit costs consisted of expenses during visit to ER of hospital for RA.
  dollars
    Inpatient visits cost | 3,089.94 (14,786.15) | 2,831.70 (14,317.53) | 1151.57 (7901.71) | 1789.30 (8142.05) | 1587.91 (9792.03) | 1309.07 (6851.41) | 1838.26 (12154.86) | 4505.60 (20528.63) | 3468.19 (15523.54) | 2353.90 (12328.42) | 1791.46 (10793.10)
    Outpatient visits costs | 4,006.13 (19,532.04) | 3,062.35 (11,564.95) | 1727.93 (3936.67) | 2263.77 (6164.69) | 1665.28 (2716.01) | 5686.02 (19928.57) | 2601.07 (11012.98) | 5363.37 (11254.35) | 4237.16 (13758.63) | 3272.09 (8075.92) | 2467.90 (8644.57)
    ER visits costs | 349.64 (1,585.83) | 328.19 (1,576.11) | 219.03 (1206.08) | 277.53 (2140.86) | 259.28 (1316.71) | 407.85 (1947.66) | 212.55 (1251.78) | 399.12 (1739.26) | 363.43 (1481.07) | 365.98 (1593.09) | 273.51 (1411.57)
All Cause Total Health Care Costs, Medical Costs, Pharmacy Costs During 12 Months Pre-Index Period [Mean (Standard Deviation); unit: dollars] — All cause total health care costs, medical costs, pharmacy costs during 12 months pre-index period are reported. All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
  dollars
    Health care costs | 24,420.92 (47,406.99) | 30,416.53 (43,264.63) | 16168.53 (25602.71) | 26501.73 (34187.93) | 17580.75 (30240.41) | 23845.95 (30481.00) | 24,401.11 (42,380.03) | 48981.85 (75040.93) | 40490.72 (57253.38) | 30609.54 (35308.08) | 21784.90 (36617.83)
    Medical costs | 19,512.32 (44,212.78) | 19,379.45 (40,053.13) | 11999.99 (22939.57) | 17366.38 (29180.07) | 12993.07 (26,623.07) | 17956.78 (26,894.74) | 17808.46 (38710.40) | 37554.08 (65360.94) | 27077.56 (48487.39) | 20335.48 (28896.19) | 15820.00 (32082.59)
    Pharmacy costs | 4,908.60 (9,860.95) | 11,037.07 (15,244.06) | 4168.54 (7951.66) | 9135.35 (13525.45) | 4587.69 (11199.66) | 5889.17 (14361.93) | 6592.65 (11444.46) | 11427.76 (33915.60) | 13413.16 (29104.61) | 10274.06 (19612.35) | 5964.90 (14230.43)
RA Related Total Health Care Costs, Medical Costs, Pharmacy Costs During 12 Months Pre-Index Period [Mean (Standard Deviation); unit: dollars] — RA related total health care costs, medical costs, pharmacy costs during 12 months pre-index period are reported. RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
  dollars
    Health care costs | 8,833.52 (25,667.44) | 14,943.61 (24,196.06) | 4546.86 (10379.97) | 9807.20 (15314.26) | 4935.77 (11793.45) | 10462.36 (22548.83) | 8151.85 (18490.62) | 15878.07 (31575.28) | 15136.67 (23086.46) | 11914.79 (20,244.11) | 7230.81 (16,844.84)
    Medical costs | 7,445.71 (25,437.86) | 6,222.23 (18,623.00) | 3098.53 (9170.64) | 4330.60 (10538.65) | 3512.47 (10696.10) | 7402.94 (21149.65) | 4651.88 (16484.62) | 10268.09 (24816.89) | 8068.79 (20919.77) | 5,991.97 (15,427.73) | 4,532.88 (14,350.99)
    Pharmacy costs | 1,215.71 (2,974.03) | 7,230.13 (13,414.82) | 1361.31 (4448.33) | 4712.28 (11103.97) | 1347.30 (4566.96) | 2272.80 (6908.41) | 2399.30 (6306.26) | 3413.49 (9249.18) | 5537.26 (11303.84) | 4,434.95 (10,153.34) | 2,211.73 (6,758.38)
Total All Cause Monthly Health Care Cost During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: dollars] — All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this baseline characteristic total all cause health care cost in dollars is reported for each month of pre-index baseline period.
  dollars
    Month 1 | 1,472.00 (3,964.00) | 1,585.23 (4,511.40) | 1,195.47 (2,995.66) | 1,268.10 (2,070.32) | 1,309.62 (3,241.11) | 1,223.86 (1,782.55) | 1,654.98 (4,444.79) | 5,422.21 (18,311.75) | 2,578.36 (9,044.31) | 1,697.90 (3,722.09) | 1,545.44 (5,285.44)
    Month 2 | 1,841.98 (5,672.40) | 1,893.55 (5,349.66) | 1,221.22 (3,437.40) | 1,302.98 (3,060.04) | 1,358.67 (4,471.99) | 1,800.75 (3,735.34) | 1,582.17 (5,171.59) | 4,457.43 (17,260.29) | 2,988.66 (8,177.26) | 1,967.35 (3,994.51) | 1,611.54 (5,610.29)
    Month 3 | 1,950.72 (6,054.56) | 1,967.88 (4,629.86) | 1,413.62 (4,763.79) | 1,991.21 (3,653.14) | 1,344.95 (4,357.56) | 1,945.43 (4,917.73) | 1,456.25 (2,597.73) | 4,999.71 (16,893.14) | 3,142.42 (6,375.80) | 2,568.07 (5,760.73) | 1,778.72 (5,905.89)
    Month 4 | 1,831.75 (6,783.17) | 2,345.62 (5,547.80) | 1,408.75 (4,353.81) | 2,483.09 (9,380.52) | 1,505.32 (6,551.42) | 2,147.16 (4,807.09) | 2,512.04 (10,555.29) | 3,173.71 (6,536.49) | 3,468.91 (9,562.43) | 2,548.52 (6,278.21) | 1,833.05 (6,224.14)
    Month 5 | 1,675.13 (6,088.40) | 3,392.53 (15,825.28) | 1,527.09 (5,071.51) | 1,758.14 (3,461.89) | 1,591.72 (5,506.24) | 2,114.46 (5,180.05) | 2,218.34 (5,995.86) | 4,185.96 (11,773.79) | 2,948.97 (6,648.21) | 2,808.88 (6,605.37) | 1,950.09 (6,657.06)
    Month 6 | 1,795.34 (5,425.88) | 2,872.44 (8,354.65) | 1,395.97 (4,745.83) | 2,739.15 (8,184.36) | 1,494.42 (3,935.51) | 2,072.51 (4,611.54) | 1,917.33 (4,986.30) | 4,055.38 (11,882.81) | 3,514.88 (8,666.83) | 2,314.86 (4,419.75) | 1,841.56 (5,579.06)
    Month 7 | 2,065.20 (5,994.05) | 2,748.68 (5,793.90) | 1,338.57 (4,608.86) | 3,155.53 (8,765.16) | 1,613.11 (4,861.36) | 2,300.37 (5,609.29) | 1,853.74 (8,578.01) | 3,973.03 (11,780.35) | 2,888.53 (7,052.99) | 3,161.07 (10,088.12) | 1,918.63 (6,333.24)
    Month 8 | 1,821.27 (5,436.36) | 2,573.90 (5,934.45) | 1,426.81 (5,137.29) | 2,851.54 (6,973.89) | 1,494.05 (6,412.22) | 1,979.07 (4,586.50) | 2,276.07 (6,439.26) | 3,345.52 (9,676.74) | 4,544.99 (15,057.51) | 2,907.13 (5,677.67) | 1,899.12 (6,435.26)
    Month 9 | 2,811.19 (11,684.53) | 2,647.26 (5,787.01) | 1,300.85 (4,397.94) | 1,799.68 (4,360.96) | 1,469.14 (5,540.05) | 2,225.15 (6,382.76) | 2,220.71 (12,367.62) | 4,008.30 (9,388.11) | 3,462.03 (9,018.17) | 2,355.49 (5,254.45) | 1,836.07 (6,502.79)
    Month 10 | 2,255.16 (10,002.22) | 2,471.86 (7,969.85) | 1,460.94 (7,614.63) | 2,441.32 (6,726.25) | 1,504.17 (6,658.33) | 2,320.68 (4,945.91) | 2,275.94 (10,695.17) | 3,353.37 (7,098.15) | 4,993.31 (21,871.26) | 2,729.46 (7,803.62) | 1,936.48 (8,342.23)
    Month 11 | 2,531.08 (10,352.92) | 2,789.28 (10,384.81) | 1,308.22 (5,002.82) | 1,584.63 (2,672.79) | 1,503.62 (4,509.59) | 1,886.96 (4,857.36) | 2,574.77 (11,572.01) | 3,795.88 (10,458.45) | 2,986.24 (7,461.79) | 2,705.38 (5,841.53) | 1,839.75 (6,472.03)
    Month 12 | 2,370.10 (10,163.97) | 3,128.29 (6,951.00) | 1,171.01 (3,347.20) | 3,126.35 (8,734.75) | 1,391.97 (4,685.03) | 1,829.55 (4,212.90) | 1,858.76 (5,981.09) | 4,211.34 (8,924.43) | 2,973.41 (7,460.54) | 2,845.43 (6,831.07) | 1,794.44 (5,550.54)
Total RA Related Monthly Health Care Cost During 12 Months Pre-Index Baseline Period [Mean (Standard Deviation); unit: dollars] — RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this baseline characteristic RA related total all cause health care cost in dollars is reported for each month of pre-index baseline period.
  dollars
    Month 1 | 406.83 (1,619.24) | 703.28 (3,907.43) | 439.11 (1,589.58) | 322.11 (844.32) | 469.85 (2,199.09) | 441.39 (1,290.59) | 539.47 (2,768.24) | 1,962.14 (13,284.62) | 430.25 (1,111.69) | 473.64 (1,356.24) | 528.95 (3,402.02)
    Month 2 | 566.83 (3,826.74) | 882.34 (4,120.86) | 469.92 (2,658.20) | 531.40 (2,601.98) | 431.85 (2,771.90) | 928.87 (3,291.21) | 549.71 (2,069.01) | 1,192.36 (7,180.33) | 1,325.06 (6,068.59) | 654.37 (1,876.46) | 578.64 (3,258.34)
    Month 3 | 655.66 (4,004.11) | 1,056.77 (3,824.32) | 454.12 (2,803.31) | 1,142.03 (3,334.59) | 456.38 (3,023.11) | 756.09 (2,747.09) | 560.10 (1,714.80) | 1,649.74 (10,509.93) | 1,020.45 (2,905.01) | 921.59 (3,769.16) | 630.44 (3,714.50)
    Month 4 | 730.91 (5,246.45) | 1,303.00 (4,313.06) | 442.85 (2,018.74) | 798.63 (2,432.86) | 482.37 (4,554.79) | 958.05 (3,302.16) | 1,202.34 (9,855.61) | 757.71 (2,576.49) | 1,277.46 (3,232.57) | 1,119.77 (4,721.57) | 662.62 (4,133.73)
    Month 5 | 685.73 (5,135.95) | 1,062.30 (2,928.13) | 486.22 (3,038.35) | 765.62 (2,130.63) | 521.77 (3,323.80) | 954.68 (3,610.34) | 1,048.93 (4,863.81) | 1,273.15 (5,820.90) | 1,164.43 (3,669.03) | 825.12 (2,359.95) | 666.50 (3,506.75)
    Month 6 | 660.86 (3,687.69) | 1,153.03 (3,383.39) | 380.78 (2,221.36) | 1,149.35 (3,733.45) | 420.73 (2,016.61) | 1,179.18 (4,190.03) | 683.35 (2,716.99) | 1,336.14 (4,584.60) | 1,512.57 (4,394.90) | 886.98 (2,654.20) | 621.82 (2,779.38)
    Month 7 | 795.24 (3,635.05) | 1,595.90 (5,028.76) | 300.98 (1,305.66) | 1,084.32 (4,484.62) | 371.06 (1,888.55) | 1,043.14 (4,077.61) | 528.57 (1,611.21) | 1,535.64 (4,984.93) | 1,580.73 (6,155.27) | 1,506.72 (8,975.05) | 643.43 (3,600.63)
    Month 8 | 684.64 (3,744.93) | 1,562.50 (5,568.83) | 354.75 (1,946.36) | 976.85 (3,453.52) | 335.36 (1,750.03) | 954.47 (3,523.14) | 860.95 (3,660.07) | 1,164.74 (4,182.09) | 1,179.40 (3,792.58) | 1,276.16 (4,023.91) | 612.85 (2,877.18)
    Month 9 | 1,146.75 (8,152.88) | 1,167.06 (2,588.52) | 323.44 (2,680.72) | 628.15 (1,892.34) | 448.58 (4,363.20) | 1,000.19 (4,066.02) | 472.76 (1,867.06) | 1,562.92 (6,092.02) | 1,152.80 (2,780.05) | 957.33 (3,882.14) | 603.72 (3,917.33)
    Month 10 | 840.51 (5,804.19) | 1,202.02 (2,951.84) | 279.40 (2,115.08) | 618.40 (1,892.74) | 248.11 (1,494.89) | 877.15 (3,123.73) | 518.84 (2,090.45) | 962.51 (3,276.90) | 2,010.47 (10,949.32) | 1,217.53 (6,154.58) | 533.13 (3,428.70)
    Month 11 | 792.87 (3,620.60) | 1,742.02 (9,856.48) | 369.35 (3,438.00) | 635.71 (1,873.22) | 321.38 (1,966.71) | 732.68 (3,025.76) | 663.43 (2,707.95) | 999.43 (3,233.47) | 1,078.26 (2,531.66) | 1,129.36 (3,563.67) | 576.61 (3,563.16)
    Month 12 | 866.68 (6,397.79) | 1,513.38 (4,866.04) | 245.94 (1,376.47) | 1,154.62 (5,835.03) | 428.33 (3,467.75) | 636.49 (1,859.90) | 523.41 (2,603.76) | 1,481.59 (4,925.66) | 1,404.77 (5,959.49) | 946.24 (3,371.70) | 572.10 (3,361.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were on Combination Therapy and Monotherapy During 90 Days After Index Date
Description: In this outcome measure number of participants who were on combination therapy with index medication and who were on monotherapy during 12 months pre-index date were reported. Participants with a use of at least 1 of 4 specific csDMARDs (methotrexate, sulfasalazine, hydroxychloroquine, leflunomide) within 90 days on or after the index date were considered as being treated with combination therapy. Participants who did not take any csDMARDs along with index medication were considered being treated with monotherapy.
Time Frame: Within 90 days after index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants
  Combination therapy | 183 | 168 | 2001 | 119 | 1373 | 266 | 279 | 194 | 101 | 350
  Monotherapy | 166 | 136 | 727 | 73 | 575 | 83 | 97 | 131 | 103 | 183

2. Primary Outcome: Number of Participants for Each of the Most Commonly Used Medications During the 12 Months Post-index Date
Description: Number of participants with most commonly used medications use during 12 months post index period are reported. The 25 most medications: 1) methotrexate sodium, 2) prednisone, 3) folic acid, 4) adalimumab, 5) etanercept, 6) acetaminophen/hydrocodone bitartrate, 7) hydroxychloroquine sulfate, 8) azithromycin, 9) levothyroxine sodium, 10) tramadol hydrochloride, 11) methylprednisolone, 12) gabapentin, 13) albuterol sulfate, 14) amoxicillin/clavulanate potassium, 15) omeprazole, 16) amoxicillin, 17) meloxicam, 18) tofacitinib citrate, 19) fluticasone propionate, 20) cyclobenzaprine hydrochloride, 21) diclofenac sodium, 22) duloxetine hydrochloride, 23) atorvastatin calcium, 24) leflunomide, 25) fluconazole. A participant could have received >=1 most common medication.
Time Frame: During 12 months post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants
  Methotrexate Sodium | 163 | 136 | 1,789 | 120 | 1,193 | 245 | 252 | 163 | 105 | 289
  Prednisone | 161 | 185 | 1,473 | 106 | 1,053 | 221 | 214 | 191 | 129 | 306
  Folic Acid | 155 | 116 | 1,616 | 109 | 1,078 | 201 | 234 | 148 | 95 | 268
  Adalimumab | 20 | 16 | 2,717 | 13 | 353 | 12 | 9 | 2 | 10 | 19
  Etanercept | 12 | 11 | 327 | 7 | 1,943 | 6 | 11 | 1 | 8 | 25
  Acetaminophen/Hydrocodone Bitartrate | 69 | 85 | 642 | 42 | 479 | 111 | 96 | 80 | 66 | 159
  Hydroxychloroquine Sulfate | 74 | 75 | 665 | 36 | 501 | 72 | 92 | 82 | 39 | 163
  Azithromycin | 75 | 87 | 621 | 33 | 447 | 76 | 89 | 78 | 44 | 151
  Levothyroxine Sodium | 70 | 56 | 508 | 34 | 369 | 64 | 75 | 61 | 44 | 124
  Tramadol Hydrochloride | 56 | 54 | 497 | 36 | 388 | 67 | 83 | 62 | 43 | 107
  Methylprednisolone | 66 | 64 | 503 | 49 | 357 | 61 | 67 | 50 | 30 | 104
  Gabapentin | 58 | 48 | 397 | 38 | 341 | 66 | 64 | 58 | 40 | 113
  Albuterol Sulfate | 56 | 59 | 433 | 25 | 321 | 50 | 53 | 53 | 35 | 99
  Amoxicillin/Clavulanate Potassium | 49 | 51 | 427 | 33 | 289 | 41 | 61 | 55 | 32 | 90
  Omeprazole | 47 | 50 | 387 | 20 | 314 | 68 | 58 | 56 | 38 | 89
  Amoxicillin | 54 | 41 | 391 | 36 | 312 | 55 | 58 | 49 | 36 | 93
  Meloxicam | 43 | 41 | 463 | 21 | 293 | 62 | 62 | 28 | 29 | 68
  Tofacitinib Citrate | 349 | 304 | 180 | 11 | 123 | 3 | 12 | 7 | 9 | 33
  Fluticasone Propionate | 47 | 49 | 322 | 25 | 269 | 62 | 56 | 45 | 26 | 83
  Cyclobenzaprine Hydrochloride | 38 | 49 | 339 | 28 | 288 | 47 | 54 | 33 | 27 | 67
  Diclofenac Sodium | 47 | 38 | 332 | 31 | 259 | 44 | 53 | 34 | 32 | 72
  Duloxetine Hydrochloride | 30 | 41 | 318 | 23 | 253 | 45 | 55 | 37 | 31 | 75
  Atorvastatin Calcium | 58 | 34 | 311 | 23 | 215 | 52 | 40 | 39 | 34 | 74
  Leflunomide | 35 | 35 | 300 | 19 | 238 | 44 | 43 | 36 | 19 | 70
  Fluconazole | 27 | 26 | 320 | 23 | 195 | 42 | 49 | 38 | 18 | 68

3. Primary Outcome: Number of Participants Who Used Opioids and Non-steroidal Anti-inflammatory Drug (NSAIDs) During 12 Months Post Index Period
Description: Number of participants who used at least 1 opioid and NSAID during post-index period are reported.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 210 | 205 | 1,623 | 104 | 1,236 | 233 | 249 | 202 | 143 | 342

4. Primary Outcome: Mean Number of Pharmacy Claims for Opioids and NSAIDS During 12 Months Post Index Period
Description: The mean number of pharmacy claims for opioids and NSAIDs during the post-index period are reported. A pharmacy claim was defined as a claim made by participants to their insurance provider in purchasing opioids and NSAIDs from the pharmacy.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 210 | 205 | 1623 | 104 | 1236 | 233 | 249 | 202 | 143 | 342
pharmacy claims | 3.68 (6.04) | 4.99 (6.87) | 3.78 (5.98) | 3.80 (6.00) | 4.13 (6.00) | 4.30 (6.04) | 4.08 (5.37) | 3.83 (5.63) | 5.19 (6.52) | 4.50 (6.23)

5. Primary Outcome: Mean Number of Days From The Index Date to the First Opioid and NSAIDs Claim During 12 Months Post Index Period
Description: Mean number of days from the index date to the first opioid and NSAIDs claim during post index period are reported.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 210 | 205 | 1623 | 104 | 1236 | 233 | 249 | 202 | 143 | 342
days
  Days to First Opioid | 85.35 (94.49) | 83.31 (95.78) | 95.67 (98.71) | 99.05 (105.20) | 94.05 (99.55) | 101.04 (102.35) | 88.81 (89.79) | 98.71 (101.38) | 81.58 (92.36) | 93.31 (96.62)
  Days to First NSAID | 116.22 (99.95) | 99.94 (95.31) | 107.03 (99.29) | 123.31 (106.32) | 105.37 (97.93) | 118.44 (107.09) | 110.65 (103.11) | 97.37 (92.35) | 92.44 (89.42) | 90.89 (93.80)

6. Primary Outcome: Number of Participants Who Used Opioids and NSAIDs While Persistent and After Persistent With Index Medication During 12 Months Post Index Period
Description: Number of participants who used opioids and NSAIDs during tofacitinib persistency and post-persistency are reported. Persistence with the index medication was defined as not having a gap in therapy of at least 60 days between fills/infusions.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants
  Used Opioids While Persistent | 138 | 128 | 1,035 | 61 | 774 | 168 | 177 | 78 | 104 | 246
  Used Opioids After Persistent | 22 | 31 | 182 | 20 | 167 | 23 | 18 | 85 | 17 | 41
  Used NSAIDs While Persistent | 94 | 85 | 769 | 43 | 535 | 100 | 122 | 39 | 60 | 146
  Used NSAIDs After Persistent | 20 | 26 | 157 | 16 | 144 | 17 | 26 | 62 | 8 | 25

7. Primary Outcome: Number of Participants Who Used Oral Corticosteroids During 12 Months Post-Index Period
Description: The number of participants who used at least 1 oral corticosteroid during the 12 months post-index period are reported.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 198 | 216 | 1,713 | 126 | 1,225 | 241 | 241 | 217 | 138 | 356

8. Primary Outcome: Number of Participants Who Were Non-persistent to Index Medication
Description: Non-persistence was defined as the gap of at least 60 days in treatment with the index medication or switching to other biologic.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 166 | 189 | 1381 | 117 | 1036 | 139 | 188 | 320 | 117 | 287

9. Primary Outcome: Number of Participants Who Switched Immediately From Index Medication
Description: Participants were classified as switched immediately if they initiated a non-index bDMARD before a 60-day gap in index medication treatment.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 41 | 70 | 575 | 33 | 451 | 49 | 55 | 3 | 34 | 112

10. Primary Outcome: Number of Participants Who Discontinued Then Restarted Index Medication
Description: Participants were classified as discontinued and then restarted index medication if there was a gap in the index therapy of at least 60 days and the first medication observed after the gap was the index medication.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 43 | 33 | 201 | 15 | 152 | 21 | 55 | 197 | 21 | 52

11. Primary Outcome: Number of Participants Who Discontinued Then Switched From Index Medication
Description: Participants were classified as discontinued and then switched from index medication if there was a gap in the index therapy of at least 60 days and the first medication observed after the gap was a bDMARD (including tofacitinib) different from index medication.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 12 | 24 | 127 | 15 | 130 | 7 | 24 | 19 | 11 | 25

12. Primary Outcome: Number of Participants Who Discontinued Without Switching or Restarting Index Medication
Description: Participants were classified as discontinued without switching or restarting index medication if they had a gap in therapy of at least 60 days and there were no claims for either the index medication or a different bDMARD for the remainder of the follow-up period.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 70 | 62 | 478 | 54 | 303 | 62 | 54 | 101 | 51 | 98

13. Primary Outcome: Number of Participants Who Switched Any Time From Index Medication
Description: Number of participants who switched from index medication to a biologic at any time during post-index period are reported.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 55 | 96 | 727 | 48 | 599 | 56 | 84 | 26 | 45 | 140

14. Primary Outcome: Number of Participants Who Re-started Index Medication at Any Time
Description: Participants who had a claim for the index medication any time after they were considered non-persistent with the index treatment (i.e, including after switching) during the 12-month follow-up are reported. Non-persistence was defined as the gap of at least 60 days in treatment with the index medication or switching to other biologic.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants | 25 | 25 | 132 | 6 | 78 | 13 | 25 | 188 | 9 | 31

15. Primary Outcome: Mean Medication Possession Ratio (MPR) for Methotrexate
Description: MPR was calculated as the total days supply of methotrexate between the first and including the last prescription/administration divided by the time between the first through and including last biologic prescription/administration days supply.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study. As per planned analysis MPR was not evaluated for Rituximab arm.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 0 | 204 | 533
ratio | 0.89 (0.16) | 0.87 (0.18) | 0.91 (0.14) | 0.92 (0.14) | 0.91 (0.14) | 0.98 (0.07) | 0.65 (0.18) |  | 0.89 (0.14) | 0.91 (0.14)

16. Primary Outcome: Proportion of Days Covered (PDC)
Description: The PDC was calculated based on total days supply over the 12 months follow-up. The PDC was calculated by using the date of service and the day supply for each fill of the index medication.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
proportion of days | 0.65 (0.32) | 0.55 (0.32) | 0.66 (0.31) | 0.56 (0.32) | 0.63 (0.32) | 0.77 (0.28) | 0.46 (0.20) | 0.63 (0.48) | 0.60 (0.31) | 0.63 (0.31)

17. Primary Outcome: Addition of Conventional Synthetic Disease-modifying Antirheumatic Drug (Cs-DMARDs) in Participants With Monotherapy
Description: Participants with monotherapy who used additional csDMARD during post index period are reported.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study. Here, "overall number of participants analyzed" signifies the participants who initiated treatment as monotherapy with index medication only.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 166 | 136 | 727 | 73 | 575 | 83 | 97 | 131 | 103 | 183
Participants | 48 | 37 | 247 | 29 | 193 | 28 | 31 | 39 | 36 | 70

18. Primary Outcome: Adherence to Cs-DMARDs in Participants With Combination Therapy
Description: Adherence was calculated as the total day supply for csDMARDs divided by the number of days from the first claim during the follow-up until the end of the follow-up.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study. Here, "overall number of participants analyzed" signifies the participants who initiated treatment as combination therapy with index medication and cs-DMARDs.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 183 | 168 | 2001 | 119 | 1373 | 266 | 279 | 194 | 101 | 350
ratio | 0.72 (0.30) | 0.79 (0.26) | 0.77 (0.27) | 0.74 (0.28) | 0.78 (0.27) | 0.79 (0.26) | 0.79 (0.27) | 0.77 (0.28) | 0.70 (0.30) | 0.80 (0.26)

19. Primary Outcome: Number of Participants Who Met Different Medication Effectiveness Criteria
Description: Adherence criteria: PDC >=0.8, proportion of days of supply during post-index period of 12 months.Dose escalation criteria: no increase in dose for index drug compared to starting dose during post-index period. Switch criteria: no switching from index drug to (different) biologic agent during post-index period. DMARD criteria: no addition of new csDMARD to index drug during post-index period. Oral glucocorticoid criteria: Participants with no claims for oral glucocorticoids in 6 months pre-index cannot receive oral glucocorticoids for greater than (>)30 days between (index date +91 days) to (index date + 365 days); or participants with claims for oral glucocorticoids in 6 months pre-index no increase in oral glucocorticoid dose during months 6-12 post-index.Injectable glucocorticoid criteria: at most 1 parenteral or intra-articular glucocorticoid joint injection on unique days after participant had been on bDMARD treatment for >3 months between (index date + 91) to (index date + 365).
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
Participants
  Met adherence criteria | 168 | 98 | 1249 | 64 | 843 | 222 | 30 | 206 | 72 | 223
  Met dose escalation criteria | 333 | 288 | 2362 | 190 | 1864 | 199 | 373 | 0 | 202 | 522
  Met switch criteria | 294 | 208 | 2001 | 144 | 1349 | 293 | 292 | 299 | 159 | 393
  Met DMARD criteria | 316 | 270 | 2458 | 165 | 1727 | 314 | 339 | 298 | 185 | 462
  Met glucocorticoid oral criteria | 285 | 240 | 2308 | 160 | 1652 | 288 | 316 | 269 | 167 | 429
  Met glucocorticoid injection criteria | 306 | 242 | 2263 | 149 | 1605 | 246 | 291 | 140 | 151 | 406

20. Primary Outcome: All Cause Inpatient Visits Costs, Outpatient Visits Costs and Emergency Room (ER) Visits Costs During 12 Months Post Index Period
Description: All cause inpatient visits costs, outpatient visits costs and emergency room visits costs during 12 months post index period are reported. Inpatient visit costs consisted of expenses during hospital visit for formal admission. Outpatient visit costs consisted of expenses when participants visited hospital but not for formal admission. Emergency room visit costs consisted of expenses during visit to hospital emergency room.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars
  Inpatient visits costs | 5,301.85 (20,548.39) | 4,326.53 (18,879.99) | 3,863.95 (20,664.73) | 4,691.74 (18,400.58) | 3,856.57 (17,506.77) | 5,260.88 (18,311.36) | 3,482.13 (15,539.56) | 11,204.53 (46,080.79) | 5,929.53 (21,129.94) | 5,995.50 (25,570.37)
  Outpatient visits costs | 11,533.02 (31,816.02) | 10,643.90 (17,097.41) | 9,477.87 (19,068.99) | 33,271.44 (38,242.58) | 10,567.29 (22,288.21) | 42,056.44 (32,134.21) | 39,161.11 (30,665.68) | 69,689.17 (66,481.44) | 28,394.20 (30,600.24) | 35,119.77 (36,208.77)
  ER visits costs | 1,330.49 (4,934.64) | 1,500.08 (3,892.48) | 1,079.34 (3,346.54) | 1,738.59 (5,234.10) | 1,176.85 (4,307.77) | 1,663.83 (4,093.45) | 1,177.78 (3,618.48) | 1,787.39 (4,392.54) | 1,567.34 (4,030.41) | 1,814.41 (6,476.07)

21. Primary Outcome: Rheumatoid Arthritis (RA) Related Inpatient Visits Costs, Outpatient Visits Costs and Emergency Room (ER) Visits Costs During 12 Months Post Index Period
Description: RA related inpatient visit costs consisted of expenses during hospital visits for formal admission for RA. Outpatient visit costs consisted of expenses when participants visited hospital but not for formal admission for RA. ER visit costs consisted of expenses during visit to ER of hospital for RA.
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars
  Inpatient visits costs | 2,465.50 (13,108.37) | 2,470.87 (13,911.22) | 2,215.74 (15,372.12) | 1,794.11 (8,062.54) | 2,054.38 (11,418.40) | 3,561.22 (14,505.62) | 2,034.70 (12,060.95) | 4,938.52 (24,124.90) | 2,143.98 (9,456.96) | 2,678.39 (15,669.24)
  Outpatient visits costs | 2,257.47 (8,687.34) | 1,773.11 (2,446.67) | 2,060.29 (5,605.48) | 3,540.19 (5,886.92) | 2,122.31 (6,842.63) | 5,412.86 (7,401.70) | 3,348.09 (6,632.70) | 9,991.58 (18,160.69) | 4,176.44 (7,257.25) | 4,166.63 (8,262.58)
  ER visits costs | 335.97 (1,902.64) | 359.62 (1,397.80) | 374.24 (1,940.56) | 351.14 (1,187.24) | 356.14 (1,979.50) | 569.19 (2,702.12) | 416.68 (1,933.80) | 403.89 (1,807.54) | 345.85 (1,771.27) | 485.19 (2,931.20)

22. Primary Outcome: All Cause Total Health Care Costs, Medical Costs, Pharmacy Costs During 12 Months Post-Index Period
Description: All cause total health care costs, medical costs, pharmacy costs during 12 months post-index period are reported. All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars
  Total health care costs | 61,431.53 (50,673.36) | 53,150.92 (35,767.69) | 66,645.17 (38,833.73) | 62,064.23 (47,099.08) | 64,120.91 (39,299.75) | 55,737.03 (42,155.65) | 58,148.31 (36,240.29) | 95,365.52 (102,623.86) | 62,120.81 (52,128.91) | 69,508.99 (48,744.63)
  Medical costs | 18,165.35 (43,146.20) | 16,470.52 (32,254.10) | 14,421.15 (32,612.17) | 39,701.78 (45,908.94) | 15,600.71 (33,988.45) | 48,981.15 (40,482.57) | 43,821.02 (36,135.48) | 82,681.09 (95,516.54) | 35,891.07 (39,557.04) | 42,929.69 (50,218.20)
  Pharmacy costs | 43,266.17 (25,298.33) | 36,680.40 (19,244.84) | 52,224.02 (23,822.84) | 22,362.45 (22,762.52) | 48,520.21 (21,330.02) | 6,755.88 (12,128.67) | 14,327.29 (21,609.36) | 12,684.43 (35,574.58) | 26,229.74 (39,070.32) | 26,579.30 (27,293.48)

23. Primary Outcome: RA Related Total Health Care Costs, Medical Costs, Pharmacy Costs During 12 Months Post-Index Period
Description: RA related total health care costs, medical costs, pharmacy costs during 12 months post-index period are reported. RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs).
Time Frame: as for outcome 2
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars
  Total health care costs | 44,134.19 (24,089.13) | 38,462.40 (22,381.48) | 54,892.62 (27,900.44) | 41,845.23 (22,687.60) | 50,531.75 (23,297.78) | 42,227.78 (34,533.34) | 43,897.47 (21,606.90) | 55,383.00 (50,554.53) | 37,868.85 (21,498.52) | 49,156.67 (31,002.05)
  Medical costs | 5,058.93 (17,558.57) | 4,603.61 (14,852.30) | 4,650.27 (17,149.92) | 5,685.44 (11,078.72) | 4,532.83 (15,083.29) | 9,543.27 (17,696.01) | 5,799.47 (14,164.57) | 15,333.99 (35,734.38) | 6,666.27 (12,568.84) | 7,330.20 (18,740.87)
  Pharmacy costs | 38,526.59 (18,005.41) | 32,697.22 (17,139.97) | 48,872.33 (22,384.60) | 17,384.65 (21,700.87) | 45,093.62 (19,352.72) | 3,679.43 (10,548.26) | 9,565.34 (17,476.03) | 3,667.78 (10,132.59) | 18,471.52 (20,373.61) | 20,603.02 (22,860.86)

24. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 1 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 1 post-index date.
Time Frame: Month 1 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 7,985.18 (5,870.38) | 6,989.92 (3,627.60) | 9,290.98 (4,894.97) | 10,394.75 (5,480.85) | 8,777.27 (5,155.60) | 8,794.60 (6,778.97) | 11,036.55 (6,382.95) | 27,231.41 (20,230.94) | 7,265.53 (7,175.27) | 10,278.66 (7,509.70)

25. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 2 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 2 post-index date.
Time Frame: Month 2 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,805.26 (8,465.89) | 3,207.83 (2,974.52) | 4,661.95 (5,512.59) | 4,734.42 (6,655.08) | 4,735.15 (7,341.43) | 4,915.29 (4,993.19) | 3,205.10 (6,755.35) | 5,169.15 (12,056.54) | 4,244.12 (6,081.42) | 4,716.32 (7,099.03)

26. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 3 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 3 post-index date.
Time Frame: Month 3 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 5,093.95 (7,838.08) | 4,551.06 (5,175.57) | 5,975.14 (6,404.19) | 6,950.34 (20,526.66) | 5,674.03 (7,388.21) | 3,047.15 (7,044.98) | 5,139.77 (6,311.03) | 5,857.31 (14,795.16) | 5,861.37 (11,900.93) | 6,395.67 (14,460.70)

27. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 4 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 4 of post-index date.
Time Frame: Month 4 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 5,079.28 (10,071.92) | 3,969.48 (5,061.60) | 5,301.22 (6,550.05) | 5,014.75 (6,964.19) | 5,120.19 (7,544.90) | 5,346.93 (11,012.15) | 4,221.26 (10,606.65) | 5,344.44 (13,741.05) | 5,977.41 (12,963.41) | 5,412.70 (5,751.93)

28. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 5 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 5 post-index date.
Time Frame: Month 5 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,122.15 (6,848.85) | 4,874.41 (9,227.40) | 4,828.27 (5,749.33) | 4,102.21 (6,198.56) | 4,915.71 (7,978.40) | 3,363.56 (5,474.43) | 5,709.69 (9,306.48) | 4,837.39 (7,827.14) | 4,489.84 (5,244.84) | 4,951.42 (6,353.78)

29. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 6 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 6 post-index date.
Time Frame: Month 6 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,867.20 (11,052.21) | 3,826.79 (6,801.85) | 5,997.83 (13,221.77) | 4,830.11 (7,660.60) | 4,982.15 (5,627.02) | 4,626.76 (8,140.63) | 3,115.80 (4,317.17) | 5,442.79 (13,221.86) | 4,359.39 (4,986.93) | 5,059.37 (5,983.06)

30. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 7 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 7 post-index date.
Time Frame: Month 7 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,950.36 (8,724.15) | 4,939.24 (11,793.47) | 5,004.78 (6,780.50) | 4,392.10 (5,205.06) | 4,817.34 (5,794.22) | 3,067.81 (4,192.17) | 4,677.76 (4,306.25) | 8,433.49 (13,389.18) | 4,465.05 (7,021.43) | 5,874.66 (10,684.51)

31. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 8 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 8 post-index date.
Time Frame: Month 8 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,815.56 (5,915.52) | 4,139.87 (6,027.39) | 5,021.37 (6,364.92) | 5,095.74 (8,352.05) | 5,068.81 (9,110.42) | 4,943.14 (7,251.38) | 3,709.37 (5,334.43) | 8,202.13 (13,851.24) | 4,886.07 (6,342.07) | 5,745.10 (8,591.42)

32. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 9 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 9 post-index date.
Time Frame: Month 9 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,300.84 (5,689.33) | 4,399.74 (7,749.58) | 5,335.04 (7,227.68) | 3,921.54 (4,739.81) | 5,210.21 (9,459.88) | 5,064.33 (9,371.11) | 5,292.97 (8,820.67) | 5,049.22 (9,633.49) | 5,716.07 (12,032.48) | 5,249.20 (8,523.88)

33. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 10 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 10 post-index date.
Time Frame: Month 10 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 5,670.69 (21,678.99) | 3,939.86 (4,973.50) | 5,186.08 (11,341.01) | 3,998.95 (5,348.32) | 4,698.56 (5,971.85) | 4,147.01 (5,145.78) | 3,975.54 (9,056.34) | 6,545.01 (14,883.32) | 3,938.69 (4,406.49) | 5,073.34 (7,324.79)

34. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 11 Post-index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 11 post-index date.
Time Frame: Month 11 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 4,244.03 (6,261.71) | 4,083.34 (7,378.37) | 5,032.88 (6,919.38) | 4,500.99 (5,936.52) | 5,202.71 (9,216.69) | 4,334.84 (6,332.45) | 4,861.39 (6,362.99) | 6,109.10 (17,250.46) | 5,248.98 (13,994.80) | 5,180.75 (6,145.81)

35. Primary Outcome: Total All Cause Monthly Health Care Cost at Month 12 Post Index Date
Description: All cause refers to cost spent due to all comorbidities including RA. Total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure total all cause health care cost in dollars is reported for Month 12 post-index date.
Time Frame: Month 12 post-index date (index date =date of first claim for index medication [bDMARDs or tofacitinib] during identification period of 3.5 years)
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 6,497.03 (16,191.59) | 4,229.36 (4,796.31) | 5,009.64 (6,414.68) | 4,128.34 (4,822.56) | 4,918.79 (7,208.45) | 4,085.60 (5,581.80) | 3,203.10 (4,275.94) | 7,144.07 (35,560.31) | 5,668.30 (12,736.72) | 5,571.79 (9,090.65)

36. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 1 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 1 post-index date.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 6,743.68 (3,290.35) | 6,021.42 (3,153.69) | 8,562.89 (4,383.18) | 9,390.90 (5,023.75) | 7,943.89 (4,187.36) | 7,850.66 (6,450.60) | 10,152.78 (5,722.77) | 22,346.69 (13,384.38) | 5,595.28 (4,234.37) | 8,937.97 (6,127.69)

37. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 2 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measurec RA related total all cause health care cost in dollars is reported for Month 2 post-index date.
Time Frame: as for outcome 25
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 2,998.35 (3,709.88) | 2,450.14 (2,559.50) | 3,876.12 (4,442.59) | 2,761.42 (2,733.37) | 3,639.87 (4,342.96) | 3,941.04 (3,879.91) | 2,102.21 (3,492.31) | 2,376.90 (8,383.96) | 2,478.72 (2,886.26) | 3,378.57 (4,598.62)

38. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 3 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 3 post-index date.
Time Frame: as for outcome 26
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,747.82 (4,128.35) | 3,494.46 (3,952.15) | 5,049.33 (5,212.08) | 3,829.80 (7,098.78) | 4,522.20 (4,443.60) | 2,108.64 (5,867.55) | 4,157.90 (5,309.22) | 2,487.38 (9,628.44) | 3,696.15 (7,327.63) | 3,987.88 (3,859.03)

39. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 4 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 4 post-index date.
Time Frame: as for outcome 27
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,935.88 (8,393.52) | 2,932.92 (4,452.72) | 4,279.35 (4,913.29) | 3,333.94 (5,238.91) | 4,058.48 (6,106.54) | 4,336.50 (10,408.87) | 2,982.49 (9,267.47) | 1,660.75 (7,016.18) | 3,209.19 (3,929.79) | 3,871.96 (3,628.35)

40. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 5 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 5 post-index date.
Time Frame: as for outcome 28
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 2,872.41 (4,212.74) | 3,192.69 (5,189.22) | 3,951.04 (4,643.52) | 2,631.47 (2,880.06) | 3,715.18 (4,674.66) | 2,408.72 (4,426.25) | 4,017.58 (4,117.99) | 2,442.36 (5,874.48) | 2,886.74 (3,679.24) | 3,430.00 (4,950.93)

41. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 6 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 6 post-index date.
Time Frame: as for outcome 29
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,914.17 (8,567.41) | 2,567.31 (3,448.98) | 4,657.35 (8,370.54) | 3,208.61 (4,754.10) | 4,017.72 (4,670.44) | 3,257.63 (4,275.02) | 2,207.60 (3,273.20) | 2,225.86 (6,782.54) | 2,848.72 (3,192.47) | 3,614.41 (4,409.61)

42. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 7 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 7 post-index date.
Time Frame: as for outcome 30
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,493.19 (3,937.61) | 3,724.00 (10,798.76) | 3,937.19 (4,482.39) | 3,091.38 (3,466.66) | 3,745.42 (4,327.50) | 2,156.48 (3,609.41) | 3,623.70 (3,763.69) | 5,701.51 (10,692.58) | 2,873.86 (5,510.48) | 3,980.53 (9,296.61)

43. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 8 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 8 post-index date.
Time Frame: as for outcome 31
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 2,724.51 (3,993.58) | 2,945.03 (5,092.32) | 4,118.25 (5,281.28) | 2,660.95 (3,160.08) | 3,837.85 (7,021.63) | 3,849.37 (5,761.95) | 2,597.10 (4,366.96) | 5,004.67 (10,146.63) | 3,122.90 (4,084.72) | 3,781.65 (5,490.15)

44. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 9 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 9 post-index date.
Time Frame: as for outcome 32
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,304.66 (4,833.81) | 2,938.67 (5,812.01) | 4,368.93 (6,456.66) | 2,782.29 (3,614.65) | 3,934.80 (4,426.58) | 3,535.00 (7,449.94) | 3,440.04 (3,674.15) | 2,618.44 (5,696.21) | 3,012.74 (4,507.57) | 3,338.46 (4,072.61)

45. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 10 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 10 post-index date.
Time Frame: as for outcome 33
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,416.78 (5,512.87) | 2,848.24 (4,237.09) | 4,146.86 (10,401.39) | 2,519.73 (3,185.01) | 3,677.71 (5,281.64) | 2,989.40 (4,049.61) | 2,972.93 (8,506.46) | 2,816.24 (7,484.20) | 2,515.85 (3,251.37) | 3,591.22 (6,160.68)

46. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 11 Post-index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 11 post-index date.
Time Frame: as for outcome 34
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,010.75 (4,511.85) | 2,418.53 (3,287.81) | 3,926.41 (4,868.49) | 2,861.97 (3,291.44) | 3,793.28 (5,725.91) | 2,982.23 (4,486.31) | 3,473.65 (3,866.51) | 3,261.20 (13,966.79) | 3,239.53 (4,890.32) | 3,588.33 (4,787.32)

47. Primary Outcome: Total RA Related Monthly Health Care Cost at Month 12 Post Index Date
Description: RA related total health care cost was calculated as the total of pharmacy cost (home healthcare cost, urgent care cost and other medical services costs) and medical cost (ambulatory cost, emergency department visits cost, inpatient admission cost and other costs). In this outcome measure RA related total all cause health care cost in dollars is reported for Month 12 post-index date.
Time Frame: as for outcome 35
Population: Analysis was performed on all participants included in the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
Number analyzed (Participants) | 349 | 304 | 2728 | 192 | 1948 | 349 | 376 | 325 | 204 | 533
dollars | 3,971.99 (7,435.02) | 2,929.00 (3,457.82) | 4,018.90 (5,462.12) | 2,772.76 (3,617.79) | 3,645.36 (4,613.68) | 2,812.13 (4,641.79) | 2,169.49 (3,163.67) | 2,441.00 (14,133.28) | 2,389.17 (2,778.68) | 3,655.69 (5,469.38)

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected and evaluated during the study
Description: Due to the nature of claims data base from which these data where queried, as planned no adverse events were collected in this study.
Arm/Group | Tofacitinib XR | Tofacitinib IR | Adalimumab | Certolizumab Pegol | Etanercept | Infliximab | Golimumab | Rituximab | Tocilizumab | Abatacept
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/49/NCT03964649/Prot_SAP_000.pdf